CLINICAL TRIAL: NCT02271841
Title: How Are Changing the Practices After the Introduction of the Pleth Variability Index? A Before/After Survey.
Status: Completed | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Patrice Forget, M.D., Ph.D., Universitair Ziekenhuis Brussel
Other Study IDs: UCLouvain
Record Dates: First submitted 2014-10-06; First posted 2014-10-22 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Fluid Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before introduction of PVI: Physicians' practices
- After introduction of PVI: Physicians' practices
  Interventions: Device: PVI

INTERVENTIONS:
Device: PVI — Pleth Variability Index
  Groups: After introduction of PVI

SUMMARY:
This study evaluated the practice before and after the introduction of a particular model pulsoxymeter giving, in addition, information on the state of fluid responsiveness of the patient.

DETAILED DESCRIPTION:
This study aims to qualify the capability of general anesthesiologist to adopt Pleth Variability Index (PVI) into their practice. It also seeks to establish whether the introduction of the PVI in the clinical practice is associated with a modification of the practice. In this scope, the intent is to see the impact of introduction of PVI monitoring on anesthesiologist practices, and to do this by comparing their survey response both before and after use of PVI in their surgeries, and to see how clinical practices for GDT and outcomes may have changed. To that end, the intent is to conduct this at sites with no current experience in use of PVI parameter, so that one can closely follow the change in clinician practice as PVI is adopted.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* ASA 1 to 3

Exclusion Criteria:

* ASA 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The plan will seek to recruit a minimum of 3 centers in Belgium and/or France who have little to no prior PVI experience, each institution requiring about a minimum of 10 participating anesthesiologists for that institution. As it may be difficult to locate a center without Masimo technology, the goal is to locate a center not actively in use with PVI technology for managing fluid responsiveness, and the clinicians are not actively consulting with Masimo
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Practice concerning fluid management | One day
  Amounts and type of fluids administered.

SECONDARY OUTCOMES:
Fluid management by center | One day
  Amounts and type of fluids administered.
Mortality after the introduction of Pleth Variability Index | 30 days after surgery
  mortality is higher in one of the two groups?

OTHER OUTCOMES:
Fluid management in the elderly person in belgium | One day
  Amounts and type of fluids administered.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium